CLINICAL TRIAL: NCT03708393
Title: Imagio Feasibility Multi-Reader, Multi-Case Study of Optoacoustic Images Versus Imagio Ultrasound to Guide Decision to Biopsy
Brief Title: Imagio Feasibility Multi-Reader, Multi-Case Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seno Medical Instruments Inc. (Industry)
Collaborators: American College of Radiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: Reader-01
Record Dates: First submitted 2018-09-28; First posted 2018-10-17 (Actual); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Intervention Model Description: This will be a controlled, blinded, multi-reader, multi-case (MRMC) study using a sequential design. The study will include 5-12 independent readers depending on qualifications and availability.
  Imagio (IUS+OA) Training to be completed prior to any reads taking place. Read 1 is immediately followed by Read 2 within the same read session.
  Read 1 (Control): Mammogram (if available) + History + IUS (stills and videos provided), IUS Probability of Malignancy (POM) and BI-RADS scored and the data form locked.
  Read 2 (Test): Mammogram (if available) + History + IUS (stills and videos provided), and Imagio (IUS+OA) (stills and videos provided). An interim IUS POM and BI-RADS is recorded as well as a combined Imagio (IUS+OA) POM and BIRADS Pre and Post SenoGram on separate data forms.
Who Masked: Outcomes Assessor
Masking Description: Independent Readers blinded to mass diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Imagio IUS (Active Comparator): Read 1 - Mammo (as available) + Imagio Ultrasound
  Interventions: Device: Imagio Ultrasound; Device: Mammography
- Imagio (IUS+OA) (Experimental): Read 2 - Mammo (as available) + (Imagio Ultrasound + OA)
  Interventions: Device: Imagio (IUS+OA); Device: Mammography

INTERVENTIONS:
Device: Imagio (IUS+OA) — The Imagio ultrasound and opto-acoustic images to be reviewed as part of the reader study
  Arms: Imagio (IUS+OA)
Device: Imagio Ultrasound — Imagio ultrasound images to be reviewed as part of the reader study
  Arms: Imagio IUS
Device: Mammography — Mammography images as available per standard of care
  Other Names: Mammo

SUMMARY:
Controlled, blinded, multi-reader, multi-case study

DETAILED DESCRIPTION:
The Imagio Feasibility Reader Study-01 Study is intended to evaluate if a subsequent pivotal study can be implemented to test prospective hypotheses for pre-specified effectiveness endpoints with an acceptable sample size. The Feasibility Study will be based on ITD masses from the PIONEER (NCT01943916) Pivotal study to simultaneously reflect the distributions with and without mammograms as well as site CDU BI-RADS scores within benign and malignant masses as strata. The study population will be split into 3 cohorts - Cohort 1, the 120 patient ITD Population used to run the primary/ secondary analyses. Cohort 2, 30 patients used to run exploratory analyses on false negative rate and Cohort 3, 5 patients used to run exploratory analyses on specific mass types

ELIGIBILITY:
Inclusion Criteria:

- Female subjects participating in the PIONEER-0 Study of the Imagio Breast Imaging System with known clinical status

Exclusion Criteria:

- Female subjects who did not have known clinical status in the PIONEER-0 Study of the Imagio Breast Imaging System with known clinical status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 155 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2018-12-09 (Actual); Study Completion 2018-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Thomas Stavros, MD, Study Director — Seno Medical
Locations (1):
- American College of Radiology, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: New Independent Reader Feasibility Study (new readers re-reading a sub-set of randomly selected images acquired during PIONEER-01 Study (NCT01943916); Reader-01 study execution dates: 13 Nov 2018 to 6 Dec 2018
Pre-assignment Details: Breast mass images were acquired during PIONEER-01 study. The Reader-01 study-single arm, sequentially read (IUS vs. Imagio [IUS+OA]), controlled, blinded, multi-reader, multi-case (MRMC) feasibility study. New readers recruited; NO new subjects were recruited. Subject baseline, demographic and safety data comes from PIONEER-01 subjects who were randomly selected for Reader-01 study. Outcome measures compared IUS vs. IUS+OA. Truth based on biopsy diagnosis or 12 Mo F/U truth panel decision.
Groups:
- Overall (Subjects Randomly Selected From PIONEER-01 Study): Each subject in all 3 cohorts had one mass that was read by all readers. Each subject served as her own control, with imaging of each mass by both IUS and IUS+OA modalities. All subjects for all 3 cohorts were included in safety analysis. All subjects for all 3 cohorts were followed and completed in the same manner. Cohort 1 (n=120 was representative of the subject population for the primary analysis, Cohort 2 (n=30) was special population for internal study of FN's and Cohort 3 (n=5) was for internal study of DCIS masses.
Period: Overall Study
Arm/Group | Overall (Subjects Randomly Selected From PIONEER-01 Study)
Started | 155
Completed | 155
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-diagnose (ITD)
Groups:
- Overall (Subjects Randomly Selected From PIONEER-01 Study): Each subject had one mass that was read by all readers. Each subject served as her own control, with imaging of each mass by both IUS and IUS+OA modalities. Therefore, baseline data are for overall population only.
Arm/Group | Overall (Subjects Randomly Selected From PIONEER-01 Study)
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 130
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 117
  More than one race | 1
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 155
Mass Diagnosis [Count of Participants; unit: Participants] — Mass diagnosis by (biopsy result or Truth Panel decision = TPB) TPB was determined as ground truth obtained during the PIONEER-01 Study.
  Participants
    Subjects: Benign (includes benign + Truth Panel Benign [TPB]) (Cohort 1) | 75
    Subjects: Malignant (Cohort 1) | 45
    Subjects: Malignant false negative in PIONEER-01 (Cohort 2) | 30
    Subjects: Malignant atypical (Cohort 3) | 5

OUTCOME MEASURES:

1. Primary Outcome: The Gain in Imagio IUS Alone Specificity vs Imagio (IUS+OA) Specificity at Fixed 95-99% Sensitivity (fSp), Cohort 1
Description: Primary effectiveness endpoint was the specificity of Imagio [IUS+OA] compared to IUS alone at fixed 95-99% sensitivity (fSp) interpolated from the area under the curve (AUC) of receiver operating characteristic (ROC) curves, averaged across all 10 independent readers. Both imaging modalities (IUS alone and IUS+OA) were read for each subject (subject as own control). Results for each imaging modality compared to biopsy diagnosis or 12-month follow-up ruling of benign as determined by truth panel (ground truth).
Time Frame: Baseline to 12 month follow-up
Population: 120 patients/masses were included in Cohort 1-the Intent-to-diagnose (ITD) population used to run the analysis to set the sample size for the future pivotal Reader-02 Study, 30 masses Cohort 2 to assess False negative rate, and 5 Cohort 3 DCIS, lymphoma, etc. masses to assess how readers scored. 155 masses in total across all cohorts analyzed for the Safety population analysis
Measure: Mean (95% Confidence Interval); unit: Percent of correct benign masses
Groups:
- IUS Alone: IUS alone imaging
- Imagio (IUS+OA): IUS+OA imaging
Arm/Group | IUS Alone | Imagio (IUS+OA)
Number analyzed (Participants) | 120 | 120
Percent of correct benign masses
  fSp (95.0%) | 80.9 [69.1 to 92.7] | 75.4 [61.5 to 89.3]
  fSp (96.0%) | 78.7 [65.7 to 91.7] | 71.4 [55.8 to 87.0]
  fSp (97.0%) | 75.8 [61.4 to 90.3] | 66.1 [48.6 to 83.7]
  fSp (97.5%) | 74 [58.7 to 89.4] | 62.8 [44.1 to 81.6]
  fSp (98.0%) | 71.8 [55.4 to 88.3] | 58.9 [38.8 to 79]
  fSp (99.0%) | 65.2 [45.8 to 84.6] | 47.7 [24.5 to 71.0]

2. Secondary Outcome: Partial Receiver Operating Characteristic (ROC) Area Under the Curve (pAUC), Cohort 1
Description: pAUC considers only the region of the ROC space that corresponds to clinically relevant values of sensitivity defined as 95% to 99% for Imagio [IUS+OA] vs. IUS alone; averaged across 10 readers.
Time Frame: Imagio [IUS+OA] and IUS readings relative to biopsy results and TRUTH PANEL review of NDU cases with follow-up at 12 months (≥11 months)
Population: Cohort 1, pAUC considers only the region of the ROC space that corresponds to clinically relevant values of sensitivity defined as 95% to 99% for Imagio [IUS+OA] vs. IUS alone; averaged across 10 readers.
Measure: Mean (95% Confidence Interval); unit: Probability as percentage
Arm/Group | Imagio IUS | Imagio (IUS+OA)
Number analyzed (Participants) | 120 | 120
Probability as percentage | 2.6 [1.9 to 3.3] | 3.0 [2.4 to 3.6]

3. Secondary Outcome: BiRads [Breast Imaging Reporting and Data System] Downgrades and Upgrades- Cohort 1
Description: The cumulative effect of downgrades and upgrades for benign masses expressed as the net gain of True Negative reads
Time Frame: Imagio [IUS+OA] and IUS readings relative to biopsy results and TRUTH PANEL review of NDU cases with follow-up at 12 months
Population: ITD Population- Number of Subjects/Masses 120
Measure: Number; unit: % of correctly identified benign masses
Arm/Group | Imagio IUS | Imagio (IUS+OA)
Number analyzed (Participants) | 120 | 120
% of correctly identified benign masses | 38.5 | 49.1

4. Secondary Outcome: The Negative Likelihood Ratio (NLR) for IUS vs. Imagio® (IUS+OA), Cohort 1
Description: NLR (Imagio [IUS+OA] vs. IUS alone); averaged across 10 readers (all readers).
Time Frame: as for outcome 2
Population: Cohort 1 - 120
Measure: Mean (99% Confidence Interval); unit: Ratio
Groups:
- IUS Alone: Results for IUS alone readings
- Imagio (IUS+OA): IUS+OA imaging
  Results for Imagio readings
Arm/Group | IUS Alone | Imagio (IUS+OA)
Number analyzed (Participants) | 120 | 120
Ratio | .049 [.04 to .07] | .094 [.08 to .11]

5. Secondary Outcome: SenoGram Usage Cohort 1 for Imagio (IUS+OA) Only
Description: SenoGram Utilization by number of readers using the SenoGram reported by the readers. SenoGram is not used for Imagio IUS Arm only Imagio (IUS+OA)
Time Frame: as for outcome 3
Population: Cohort 1
Measure: Number; unit: participants
Arm/Group | Imagio IUS | Imagio (IUS+OA)
Number analyzed (Participants) | 120 | 120
participants | NA — SenoGram is not used for Imagio IUS Arm only Imagio (IUS+OA) | 111

6. Secondary Outcome: SenoGram Performance
Description: Sensitivity of SenoGram estimated from cross-validation - Cohort 1
Time Frame: as for outcome 3
Population: ITD Population
Measure: Number; unit: Percent
Arm/Group | Imagio IUS | Imagio (IUS+OA)
Number analyzed (Participants) | 120 | 120
Percent | NA — SenoGram not used for IUS Arm | 98.0

7. Secondary Outcome: SenoGram Performance
Description: Specificity of SenoGram estimated from cross-validation
Time Frame: as for outcome 3
Population: ITD Population - Cohort 1
Measure: Number; unit: Percent
Arm/Group | IUS Alone | Imagio (IUS+OA)
Number analyzed (Participants) | 120 | 120
Percent | NA — SenoGram not used for IUS Arm | 62.2

ADVERSE EVENTS:
Time Frame: Baseline to 12 months +/- 30 days follow-up. Adverse Events were recorded from the use of the Imagio during the original PIONEER Study and reported out for those participants/masses selected for the Reader-01 Independent Reader Study.
Groups:
- Overall (Masses Randomly Selected From PIONEER-01 Study): Each subject had one mass that was read by all readers. Each subject served as her own control, with imaging of each mass by both IUS and IUS+OA modalities. Therefore, safety data are for overall population only.
Arm/Group | Overall (Masses Randomly Selected From PIONEER-01 Study)
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 0/155
Other Adverse Events (participants affected / at risk) | 0/155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03708393/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT03708393/SAP_001.pdf